CLINICAL TRIAL: NCT03273296
Title: Effect of Antibiotics on Gut Microbiome and Plasma Metabolome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: University of California, San Diego (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1341/6.00.00/2017
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Microbial Colonization
Keywords: microbiota; metabolize
MeSH Terms: conditions — Communicable Diseases | interventions — Amoxicillin; Azithromycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Amoxicillin (Active Comparator)
  Interventions: Drug: Amoxicillin
- Azithromycin (Active Comparator)
  Interventions: Drug: Azithromycin
- Vancomycin (Active Comparator)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin (po) 500 mg x 3 per day for 3 days.
  Arms: Amoxicillin
Drug: Azithromycin — Azithromycin (po) 500 mg x 1 on day 1, 250 mg x 1 on day 2, and 250 mg x 1 on day 3.
  Arms: Azithromycin
Drug: Vancomycin — Vancomycin (po) 125 mg x 4 per day for 3 days.
  Arms: Vancomycin

SUMMARY:
In recent years it has been observed that the gut microbiome can produce metabolites into systemic circulation and thus have important health effects even outside the gastrointestinal system. These metabolites may play a role in the pathogenesis of common public health problems such as diabetes, obesity and cardiovascular disorders. Modern techniques of mass spectrometry-based metabolomics from peripheral blood and gut metagenome sequencing now enable detailed examination of these processes. Using samples from the FINRISK 2002 cohort, collected by the National Institute for Health and Welfare, we are currently determining the gut microbiome and plasma metabolome from > 7000 participants with 15 years of follow-up for various health outcomes. This is one of the largest materials of its kind world-wide. The design does not, however, allow us to draw causal conclusions on the roles of gut bacteria in the composition of plasma metabolome. To enable conclusions which go beyond statistical associations, we now propose an extension to the FINRISK 2002 study, where we alter the gut bacteriome with a short course of antibiotics and then examine whether a change in plasma metabolomics profile will follow. At the same time the trial will give important novel information about the effects of commonly used antibiotics on gut bacteriome and on general health.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in the FINRISK 2002 survey and current residence in Helsinki metropolitan area.
* Age range 40-74 years among men and 50-74 years among women.

Exclusion Criteria:

* Known allergy to any antibiotic
* A course of antibiotic during the past year
* Acute infection
* Any major illness (history of myocardial infarction, stroke, diabetes, liver or kidney disease, cancer, psychiatric disease). Uncomplicated hypertension is allowed. Likewise, statin treatment and women's hormone replacement therapy are allowed.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Microbiome | Baseline: 0 days; repeat assessments 2 days and 28 days after end of antibiotics.
  Change in gut microbiome from baseline to repeat assessments.
Metabolome | Baseline: 0 days; repeat assessments 2 days and 28 days after end of antibiotics.
  Change in circulating metabolome from baseline to repeat assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Aki Havulinna, MD, PhD, Principal Investigator — Finnish Institute for Health and Welfare; Markus Perola, DSc (tech.), Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- Finnish Institute for Health and Welfare, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes